CLINICAL TRIAL: NCT05334706
Title: A Non-Randomized, Open-Label Study to Assess the Reduction of Human Papillomavirus (HPV) Viral Infectivity and Transmission in HPV16/18-Positive Women After Vaccination With 9vHPV, a Multivalent L1 Virus-like Particle Vaccine, Evaluated in Cervical, Anal and Oral Samples Obtained After One, Two, and Three Vaccine Doses (RIFT-HPV1/RIFT-HPV2)
Brief Title: A Study to Assess the Reduction of Human Papillomavirus (HPV) Viral Infectivity and Transmission in HPV-Positive Women After Vaccination With 9vHPV (RIFT-HPV)
Acronym: RIFT-HPV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miquel Angel Pavon Ribas (Other)
Collaborators: Hospital del Mar (Other); Catalan Institute of Health (Other Government)
Responsible Party: Sponsor-Investigator, Miquel Angel Pavon Ribas, Head of the Laboratory of Infections and Cancer (INCALAB)., Institut d'Investigació Biomèdica de Bellvitge
Organization: Institut d'Investigació Biomèdica de Bellvitge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIFT-HPV; 2021-005229-26 (EudraCT Number)
Record Dates: First submitted 2022-04-05; First posted 2022-04-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cervical Intraepithelial Neoplasia Grade I/ II/ III (CIN I/II/III); Human Papillomavirus (HPV) Infections; High-risk HPV; HPV-16/ 18
Keywords: Cervical cancer; Cervical Intraepithelial Neoplasia Grade I/ II/ III (CIN I/II/III); Squamous Intraepithelial Lesions of the Cervix, High/ Low Grade.; Uterine Cervical Neoplasms; Human Papillomavirus (HPV) Infections; High-risk HPV; HPV-16/ 18; HPV DNA Tests; Anyplex HPV28; HPV Vaccines; HPV Nonavalent Vaccine; Gardasil-9; 9vHPV; cLIA; HaCaT Cells; Keratinocytes; Cell Culture; ELISA; Immunoassay; Electron Microscopy
MeSH Terms: conditions — Papillomavirus Infections; Infections; Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions of the Cervix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaccination (Experimental): Single arm, vaccination with 9vHPV in a 3-dose regimen (Day 1, Month 2, Month 6).
  Interventions: Biological: Nonavalent HPV vaccine (9vHPV/Gardasil-9™).

INTERVENTIONS:
Biological: Nonavalent HPV vaccine (9vHPV/Gardasil-9™). — Sterile suspension, 0.5 ml dose, intramuscular administration in a 3 dose-regimen (Day 1, Month 2, Month 6), prepared from the highly purified virus-like particles (VLPs) of the major capsid L1 protein from 9 HPV types: 6/11/16/18/31/33/45/52/58.
  9vHPV is currently indicated in the EU in individuals from 9 years of age for the prevention of diseases caused by vaccine's 9 HPV types: genital warts (HPV6 and 11) and premalignant lesions and cancers affecting the cervix, vulva, vagina and anus (HPV16, 18, 31, 22, 45, 52 and 58). It was authorized for marketing in the EU on June 9th, 2015.

SUMMARY:
This is a non-randomized, open label study to assess the reduction of Human Papillomavirus (HPV) infectivity and transmission in women positive for HPV16 and/or 18 in a cervical, oral and anal sample and vaccinated with 9vHPV/Gardasil-9™.

The primary objective of the study is to demonstrate that vaccination with a 3-dose regimen of 9vHPV will reduce viral infectivity in HPV 16/18/16+18-positive women. This objective rests upon the hypothesis that, since vaccination with 9vHPV triggers the production of type-specific HPV antibodies which are exudated to the cervical and other infected mucosae, these antibodies adhere to and neutralize newly produced HPV 16/18 viral particles also present in the mucosae, thus reducing HPV's infective capacity and transmission to sexual partners.

Secondary objectives of the study are:

* To determine HPV antibody levels before and after vaccination for each of the 9vHPV-covered HPV types (6, 11, 16, 18, 31, 33, 45, 52, and 58), to distinguish an induced antibody production due to 9vHPV vaccination from a natural response to an HPV infection (when antibody production is expected to be lower).
* To demonstrate viral infectivity reduction in HPV 16/18/16+18 after vaccination with 1-dose or 2-dose regimen of 9vHPV. Since antibody production after administration of 2 vaccine doses is not inferior to 3 doses, infectivity reduction is expected to be detected after 2 doses, and at least partially after one dose.

The main endpoint of the study is the evaluation of the HPV infective capacity in cervical, anal and oral samples from HPV 16, 18 or 16+18-positive women, using a cellular assay that models in-vitro the cervical mucosa. In brief, the specific HPV biomarker E1^E4 is measured in HaCaT keratinocytes after being cultured with study samples and thus, exposed to HPV16/18 viral particles. A reduction in E1^E4 expression is expected for keratinocytes exposed to samples taken after vaccination with 9vHPV, since the specific HPV antibodies also present in these samples would bind HPV viral particles and prevent infection of cultured keratinocytes.

Other endpoints included in the study are:

* Detection of antibodies against HPV types covered by 9vHPV (6/11/16/18/31/33/45/52/58) by specific immunoassays (ELISA, cLIA).
* HPV16/18 virion detection using ELISA and electronic microscopy.
* HPV DNA detection and genotyping, using Anyplex HPV28. These endpoints are performed in cervical, anal and oral samples from HPV 16, 18 or 16+18-positive women
* Titration of antibodies against HPV types covered by 9vHPV in serum samples from HPV 16, 18 or 16+18-positive women using ELISA or cLIA.

A minimum of 39 and 30 women will be enrolled in two different study population cohorts, respectively:

* RIFT-HPV 1 cohort: non-vaccinated adult women aged 35 years or older, positive for HPV16-, 18-, or double positive for 16 and 18, without lesion or with cervical intraepithelial neoplasia (CIN) 1/2 lesion eligible for conservative treatment.
* RIFT-HPV 2 cohort: non-vaccinated adult women aged 27 years or older, positive for HPV16-, 18-, or double positive for 16 and 18, with multiple cervical, vulvar and/or anal lesions, with cervical lesions eligible for conservative treatment.

Candidates to participate in the study are selected according to the HPV DNA test result in a cervical sample taken in their routine cervical cancer screening visit or in their routine gynaecological follow-up visit.

There is no control group in this study: all participants are expected to complete all the per-protocol procedures in a total of 4 study visits within an average of 7 months' duration: Visit 1/ Day1, Visit 2/Month 2, Visit 3/Month 6, and Visit 4/Month 7.

The study procedures are the following:

* Pregnancy test on a urine sample in Visit 1 (pregnant women are excluded from the study).
* Completion of a questionnaire about the participant's health status, use of oral contraception and sexual activity in Visits 1 and 4.
* Cervical, anal oral and blood sample collection Visits 1, 2 and 3 before receiving 9vHPV vaccination, and in Visit 4.
* Intramuscular administration of 9vHPV in a three-dose regimen in Visits 1, 2 and 3.

Regarding data analysis for primary objective assessment, differences in the infectivity rate before (Day 1/ Visit 1) and after vaccination with 3 doses of 9vHPV (Month 7/ Visit 4) will be compared in cervical, anal and oral samples using non-parametric Wilcoxon signed rank test. The same assessment will be done in 1- or 2-dose vaccination scenario.

Antibody production before and after vaccination will be summarized for each of the 9vHPV-covered HPV types.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* Aged 35 or 27 years or older for RIFT-HPV Cohort 1 and 2 respectively, attending a routine cervical cancer screening visit or gynaecological visit.
* Positive for HPV16, 18 or double-positive for 16 and 18 and negative for the rest of high-risk HPV types in a cervical sample.
* Recently diagnosed for their HPV-positivity (within the last 24 months).
* Meet one of the following criteria:

have no apparent cervical lesion (Cohort 1). have a CIN1/2 lesion which is eligible for conservative treatment (cohort 1). have multiple cervical, vulvar and/or anal lesions, and cervical lesions are eligible for conservative treatment (Cohort 2).

Exclusion Criteria:

* Presence of any cervical lesion that requires clinical intervention within 7 months that could significantly affect cervical epithelia (and therefore, HPV viral production), such as cervical conization.
* History of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention.
* History of allergy to any vaccine component, including aluminum, yeast, or BENZONASETM (nuclease, Nicomedia).
* History of thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection of study vaccine.
* History of splenectomy.
* History of ano-genital cancer or HPV-related head and neck cancer.
* Pregnancy at the time of signing informed consent or planning to become pregnant within the full duration of the study.

Min Age: 27 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Rift-HPV 1 Cohort: Non-vaccinated, HPV16-, HPV18- or 16 and 18-positive adult women (35 years or older) attending routine cervical cancer screening or the gynaecology unit.
  Rift-HPV 2 Cohort: Non-vaccinated, HPV16-, HPV18- or 16 and 18-positive adult women (27 years or older) with multiple cervical, vulvar and/or anal lesion attending the gynaecology unit.
Enrollment: 69 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that vaccination with a 3-dose regimen of 9vHPV will change viral infectivity in cervical, anal and oral samples from HPV 16/18/16+18-positive women. | 7 month
  In-vitro infectivity evaluation of cervical, anal, and oral samples collected before and after 9vHPV vaccination, by expression of E1^E4 HPV biomarker in HaCaT keratinocytes.
Detection of HPV 6/11/16/18/31/33/45/52/58 L1 antibodies in cervical, anal and oral samples collected before and after 9vHPV vaccination, using ELISA and cLIA. | 7 month
  This endpoint will allow to associate the reduction in viral infectivity with the presence of neutralizing antibodies.
HPV16/18 virion detection in cervical, anal and oral samples collected before and after 9vHPV vaccination. | 7 month
  HPV16/18 virion detection will be carried out using ELISA and electronic microscopy in cervical, anal and oral samples collected before and after 9vHPV vaccination.
HPV DNA detection in cervical, anal and oral samples collected before and after 9vHPV vaccination. | 7 month
  HPV DNA detection will be performed using Anyplex HPV28 in cervical, anal and oral samples collected before and after 9vHPV vaccination.
HPV DNA genotyping in cervical, anal and oral samples collected before and after 9vHPV vaccination. | 7 month
  HPV DNA genotyping will be performed using Anyplex HPV28 in cervical, anal and oral samples collected before and after 9vHPV vaccination.

SECONDARY OUTCOMES:
To determine HPV antibody titration before and after vaccination for each of the 9vHPV-covered HPV types (6, 11, 16, 18, 31, 33, 45, 52, and 58). | 7 month
  To determine HPV 6/11/16/18/31/33/45/52/58 L1 antibody titration in serum samples collected before and after 9vHPV vaccination, using ELISA for types 16 and 18 in samples from RIFT-HPV 1 and 2 study cohorts, using cLIA for all 9vHPV-covered types except 16 and 18, in samples from RIFT-HPV 1 study cohort.
To demonstrate viral infectivity change in cervical, oral and anal samples from HPV 16/18/16+18-positive women after vaccination with 1-dose or 2-dose regimen of 9vHPV. | 7 month
  In-vitro infectivity evaluation of cervical, anal, and oral samples collected before and after 9vHPV vaccination with 1st dose and 2nd dose, by expression of E1^E4 HPV biomarker in HaCaT keratinocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Eulàlia Fernández Montolí, PhD - MD, Principal Investigator — Gynaecology Unit, Bellvitge University Hospital (HUB), L'Hospitalet del Llobregat, Spain.; Francesc Xavier Bosch José, PhD - MD, Principal Investigator — Cancer Epidemiology Research Program (PREC), Catalan Institute of Oncology (ICO-Hospitalet)/Bellvitge Biomedical Research Institute (IDIBELL), L'Hospitalet de Llobregat, Spain.
Locations (1):
- Gynaecology Unit, Bellvitge University Hospital (HUB), L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosch FX, Broker TR, Forman D, Moscicki AB, Gillison ML, Doorbar J, Stern PL, Stanley M, Arbyn M, Poljak M, Cuzick J, Castle PE, Schiller JT, Markowitz LE, Fisher WA, Canfell K, Denny LA, Franco EL, Steben M, Kane MA, Schiffman M, Meijer CJ, Sankaranarayanan R, Castellsague X, Kim JJ, Brotons M, Alemany L, Albero G, Diaz M, de Sanjose S; ICO Monograph 'Comprehensive Control of HPV Infections and Related Diseases' Vaccine Volume 30, Supplement 5, 2012. Comprehensive control of human papillomavirus infections and related diseases. Vaccine. 2013 Dec 30;31 Suppl 6:G1-31. doi: 10.1016/j.vaccine.2013.10.002. PMID 24331817
- [Background] Schiffman M, Doorbar J, Wentzensen N, de Sanjose S, Fakhry C, Monk BJ, Stanley MA, Franceschi S. Carcinogenic human papillomavirus infection. Nat Rev Dis Primers. 2016 Dec 1;2:16086. doi: 10.1038/nrdp.2016.86. PMID 27905473
- [Background] Castle PE, Rodriguez AC, Bowman FP, Herrero R, Schiffman M, Bratti MC, Morera LA, Schust D, Crowley-Nowick P, Hildesheim A. Comparison of ophthalmic sponges for measurements of immune markers from cervical secretions. Clin Diagn Lab Immunol. 2004 Mar;11(2):399-405. doi: 10.1128/cdli.11.2.399-405.2004. PMID 15013994
- [Background] Schwarz TF, Kocken M, Petaja T, Einstein MH, Spaczynski M, Louwers JA, Pedersen C, Levin M, Zahaf T, Poncelet S, Hardt K, Descamps D, Dubin G. Correlation between levels of human papillomavirus (HPV)-16 and 18 antibodies in serum and cervicovaginal secretions in girls and women vaccinated with the HPV-16/18 AS04-adjuvanted vaccine. Hum Vaccin. 2010 Dec;6(12):1054-61. doi: 10.4161/hv.6.12.13399. Epub 2010 Dec 1. PMID 21157180
- [Background] Parker KH, Kemp TJ, Pan Y, Yang Z, Giuliano AR, Pinto LA. Evaluation of HPV-16 and HPV-18 specific antibody measurements in saliva collected in oral rinses and merocel(R) sponges. Vaccine. 2018 May 3;36(19):2705-2711. doi: 10.1016/j.vaccine.2018.03.034. Epub 2018 Apr 6. PMID 29631883
- [Background] Dillner L, Bekassy Z, Jonsson N, Moreno-Lopez J, Blomberg J. Detection of IgA antibodies against human papillomavirus in cervical secretions from patients with cervical intraepithelial neoplasia. Int J Cancer. 1989 Jan 15;43(1):36-40. doi: 10.1002/ijc.2910430109. PMID 2536005
- [Background] Wang Z, Hansson BG, Forslund O, Dillner L, Sapp M, Schiller JT, Bjerre B, Dillner J. Cervical mucus antibodies against human papillomavirus type 16, 18, and 33 capsids in relation to presence of viral DNA. J Clin Microbiol. 1996 Dec;34(12):3056-62. doi: 10.1128/jcm.34.12.3056-3062.1996. PMID 8940448
- [Background] Cameron JE, Snowhite IV, Chaturvedi AK, Hagensee ME. Human papillomavirus-specific antibody status in oral fluids modestly reflects serum status in human immunodeficiency virus-positive individuals. Clin Diagn Lab Immunol. 2003 May;10(3):431-8. doi: 10.1128/cdli.10.3.431-438.2003. PMID 12738644
- [Background] MacCosham A, El-Zein M, Burchell AN, Tellier PP, Coutlee F, Franco EL. Transmission reduction and prevention with HPV vaccination (TRAP-HPV) study protocol: a randomised controlled trial of the efficacy of HPV vaccination in preventing transmission of HPV infection in heterosexual couples. BMJ Open. 2020 Aug 11;10(8):e039383. doi: 10.1136/bmjopen-2020-039383. PMID 32788190
- [Background] Ozbun MA. Infectious human papillomavirus type 31b: purification and infection of an immortalized human keratinocyte cell line. J Gen Virol. 2002 Nov;83(Pt 11):2753-2763. doi: 10.1099/0022-1317-83-11-2753. PMID 12388811
- [Derived] Lopez-Codony V, de Andres-Pablo A, Ferrando-Diez A, Fernandez-Montoli ME, Lopez-Querol M, Tous S, Ortega-Exposito C, Torrejon-Becerra JC, Perez Y, Ferrer-Artola A, Sole-Sedeno JM, Grau C, Ruperez B, Saumoy M, Sanchez M, Peremiquel-Trillas P, Bruni L, Alemany L, Bosch FX, Pavon MA. Assessing the reduction of viral infectivity in HPV16/18-positive women after one, two, and three doses of Gardasil-9 (RIFT): Study protocol. PLoS One. 2024 May 20;19(5):e0304080. doi: 10.1371/journal.pone.0304080. eCollection 2024. PMID 38768231
- See also: Transmission Reduction and Prevention with HPV Vaccination (TRAP-HPV) Study: A Randomized Controlled Trial of the Efficacy of HPV Vaccination in Preventing Transmission of HPV Infection in Heterosexual Couples. — https://clinicaltrials.gov/ct2/show/study/NCT01824537